CLINICAL TRIAL: NCT05519917
Title: An Open-label, Single-arm, Interventional Clinical Study to Evaluate the Efficacy of Afatinib in Skull Base Chordoma
Brief Title: Study to Evaluate the Efficacy of Afatinib in Skull Base Chordoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-610
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Chordoma of Clivus
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Afatinib (Experimental): Subject meeting the inclusion criteria will take afatinib (40 mg daily) orally, 4 weeks for a cycle.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Subjects will receive evaluations at the beginning of treatment, after every three cycles and at the end of the whole study.

SUMMARY:
This is a single arm, open label, single center, and prospective, interventional study to explore clinical efficacy of afatinib in patients with chordoma of skull base. Subject meeting the inclusion criteria will take afatinib (40 mg daily) orally, 4 weeks for a cycle. The primary objective is to assess the efficacy of afatinib in chordoma of skull base by objective response rate (ORR). The Secondary objectives is to assess progression free survival (PFS), overall survival (OS), tumor response duration and tumor shrinkage degree in patients with chordoma of skull base after using afatinib; to evaluate the safety and tolerability of afatinib in patients with chordoma of skull base.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years and above;
* Patients with pathologically proven EGFR and/or HER2 expressing relapsed or residual chordoma of skull base, inappropriate or unwilling to receive surgery or radiotherapy;
* Adequate bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 75 x 109/L);
* An adequate renal function with GFR ≥ 45 ml/min calculated by Cockroft-Gault formula;
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ 3 times ULN;
* Ability to swallow medication;
* Able to understand and provide written informed consent prior to any study procedures.

Exclusion Criteria:

* Life expectancy of less than 3 months;
* Known hypersensitivity to afatinib;
* Major surgery less than 4 weeks prior to start of the study;
* Patients who once participated in other clinical trials within 14 days before the initiation of the study;
* Systemic anti-cancer therapy within 28 days prior to start of the study;
* No tumor progression after radiation therapy prior to start of the study;
* History or presence of serious cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia, and myocardial infarction within 6 months prior to inclusion;
* Known pre-existing interstitial lung disease;
* No response after 2-week active treatment for known CTCAE Grade 3 or Grade 2 rash/acne;
* Any history or presence of poorly controlled gastrointestinal disorders that may worsen after administration and could affect the absorption of the study drug (e.g. diarrhea, Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption);
* Active hepatitis B infection (HepB sAg and/ or Hep B DNA positive), active hepatitis C infection (Hep C RNA positive), active tuberculosis and/or known HIV carrier;
* Using other drugs that may influence afatinib and cannot be discontinued during the study, including but not limited to:
* Potent P-gp inhibitors: including but not limited to ritonavir, cyclosporine A, ketoconazole, itraconazole, erythromycin, verapamil, quinidine, tacrolimus, nelfinavir, saquinavir and amiodarone);
* Potent P-gp inducers: including but not limited to rifampin, carbamazepine, phenytoin, phenobarbital or St. John's wort).
* Pregnant or lactating women;
* Other invasive malignancies diagnosed within the last 5 years (except non-melanoma skin cancer and localized cured prostate and cervical cancer);
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months after enrollment
  Proportion of patients with reduction in tumor volume to a predefined value for a minimum period. Generally, ORR is defined as the sum of complete response and partial response. The best response, that is, the best response throughout the study, will be evaluated.

SECONDARY OUTCOMES:
Progression-free survival | 12 months after enrollment
  duration from the date of inclusion until the date of objective tumor progression or death.
Overall survival | 12 months after enrollment
  duration from the date of inclusion until the date of death.
Duration of response | 12 months after enrollment
  duration of partial response and complete response, that is, duration from effective date to the date of proved tumor progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No